CLINICAL TRIAL: NCT04375904
Title: 'SOURCE - LUNG' Stereotactic Ablative Radiation Therapy Of UltRaCEntral LUNG Tumours
Brief Title: 'SOURCE - LUNG' Stereotactic Ablative Radiation Therapy Of UltRaCEntral LUNG Tumours (SOURCE Lung)
Acronym: SOURCE Lung
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Trials Ireland (Network)
Collaborators: Technological University Dublin (Unknown); University College Dublin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTRIAL-IE 18-33
Record Dates: First submitted 2020-04-23; First posted 2020-05-06 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: NSCLC/Oligometastatic Cancer (Single Lung Lesion)
Keywords: Lung cancer; Non-small cell lung cancer; Ultracentral; Stereotactic ablative radiation therapy; Oligometastatic cancer; Single lung lesion
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a phase II non-randomised, multi-centre, single arm trial assessing the safety of patients receiving image guided SABR in 8 fractions of 7.5Gy. The treatment will adhere to organ at risk dose-volume histogram constraints allowing a minimum dose coverage of 75% to 95% of the planning target volume (PTV) coverage, and a minimum dose of 75% to 99% of the gross tumour volume (GTV), using dose intensity modulation. These minimums are chosen to represent at least an equivalent BED to the RT standard fractionation of 55 Gy in 20 fractions based on actual treatment dose of 7.5 Gy in 8 fractions. The safety of the regimen will be based on the rate of ≥ Grade 3 treatment related toxicities per CTCAE V5 occurring between start of treatment and one-year from the end of treatment, which are possibly, probably or definitely related to radiotherapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Radiation (Experimental): Treatment will be delivered via image-guided (IG)-SABR in 8 fractions of 7.5Gy. OAR constraints must be respected but minimum dose coverage of 75% to 95% of the PTV will be allowed and minimum dose of 75% to 99% of the GTV will be allowed. The minimums are chosen to represent at least an equivalent BED to the RT standard fractionation of 55 Gy in 20 fractions based on actual treatment dose of 7.5Gy in 8 fractions. A total of 60 evaluable patients will be required for the study. The sample size was calculated using continuous monitoring for toxicity, up to one year post RT, using a Pocock-type boundary. Accrual will be halted if excessive numbers of ≥ Grade 3 TxR-AEs are seen. The regime will not be considered to be safe if >25% of evaluable patients experience a ≥ Grade 3 treatment-related adverse event (TxR-AE) by the end of 1-year post-RT. This study will be considered adequately safe if ≤ 25% of evaluable patients experience ≥ Grade 3 TxR-AE by the end of 1 year post-RT.
  Interventions: Radiation: Image-Guided Stereotactic Ablative Radiotherapy (IG-SABR)

INTERVENTIONS:
Radiation: Image-Guided Stereotactic Ablative Radiotherapy (IG-SABR) — Image-Guided Stereotactic Ablative Radiotherapy (IG-SABR) delivered in 8 fractions of 7.5 Gy. OAR constraints must be respected but a minimum dose coverage to 95% of the PTV will be allowed down to 75% and a minimum dose to 99% of the GTV allowed at 75%. Respiratory monitoring/active respiratory management will be used. Plans will be created and delivered using photon beams with energies between 6-10 MV.

SUMMARY:
This is a phase II, non-randomised study examining the safety of treating high risk centrally located non-small cell lung cancer (NSCLC) tumours and single pulmonary oligometastatic lesions using radiation therapy (RT), for patients whose disease is inoperable. The method of delivering the RT in this study is image guided stereotactic ablative radiation therapy (IG-SABR). This method involves using imaging to ensure the radiation is being delivered to the correct location within the body and using higher than normal doses per treatment (fraction) to treat the lung cancer (NSCLC)/oligometastatic lung lesion. This study aims to determine its safety by looking at the number and severity of side effects. This study will deliver 8 treatments/fractions of RT with 7.5 Gy delivered in each fraction. To be eligible for this study the initial treatment plan for the patient must be shown to not fulfil certain criteria relating to doses to the tumour and surrounding normal tissue. This study has its own study specific criteria which must be adhered to. Translational sub-studies (optional) are open to patients in participating centres only. Patients will have the option to consent to participating in both translational studies or to neither.

DETAILED DESCRIPTION:
This study is a phase II non-randomised, multi-centre, single arm trial of image-guided (IG)-SABR for patients with high-risk centrally located T1-T4 lung tumours (NSCLC) or a single pulmonary oligometastatic lesions. Treatment will consist of IG-SABR using a total of 8 fractions of 7.5 Gy per fraction adhering to organ at risk dose-volume histogram constraints allowing a minimum dose coverage of 75% to 95% of the planning target volume (PTV) coverage, and a minimum dose of 87% to 99% of the gross tumour volume (GTV), using dose intensity modulation.

The primary aim of the study is to determine the safety of the 8 x 7.5 Gy treatment regimen on the basis of the rate of ≥ Grade 3 treatment related toxicity using NCI CTCAE V5, in patients with medically inoperable early stage, ultracentrally located lung tumours. This is defined by central tumours which are not fulfilling the conservative hybrid DVCs of the LungTech (Adebahr et al., 2015), RTOG 0813 (Bezjak et al., 2015) studies and current UK consortium guidelines with full dose coverage, but which subsequently meet SOURCE DVC's with potentially reduced dose coverage. To remain in line with international practice, the SOURCE Lung protocol was amended to reduce near maximum dose constraints to 0.1cc for OARs (Diez et al. 2022). Toxicities occurring between start of treatment and one-year from the end of treatment, which are possibly, probably or definitely related to radiotherapy will be assessed.

A total of 60 evaluable patients will be required for the study. The sample size was calculated using continuous monitoring for toxicity, up to one year post RT, using a Pocock-type boundary. Accrual will be halted if excessive numbers of ≥ Grade 3 TxR-AEs are seen. The regime will not be considered to be safe if >25% of evaluable patients experience a ≥ Grade 3 treatment-related adverse event (TxR-AE) by the end of 1-year post-RT. This study will be considered adequately safe if ≤ 25% of evaluable patients experience ≥ Grade 3 TxR-AE by the end of 1 year post-RT.

The enrolment period is expected to be 6 years.

Toxicity assessments will be carried out weekly during radiotherapy (RT), at 2, 4 and 8-weeks post-treatment and at 3, 6, 9, 12, 18, 24 months post treatment and annually thereafter to 5 years post treatment.

Translational Sub-Study 1 (Raman spectroscopic analysis) - Primary aim is to undertake biomarker discovery using label-free Raman spectroscopy coupled with multivariate statistical methods to identify spectral biomarkers that could:

1. Predict response based on individual radiation sensitivity
2. Monitor response based on individual radiation sensitivity

Translational Sub-Study 2 (Proteomic analysis) - Primary aim is to use proteomic analysis of sequential blood samples before, during and after treatment to detect changes in protein expression profiles that may predict outcome and identify prognostic biochemical markers of early toxicity.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent obtained prior to any study-specific procedures
2. ≥ 18 years of age
3. Life expectancy >6 months
4. ECOG (Eastern Cooperative Oncology Group) performance status 0-2
5. Histological diagnosis (biopsy or cytology) or radiological diagnosis (PET-positive FDG-avid tumour which has only one lesion to be treated for the purpose of the study / CT-based diagnosis for non FDG-avid tumour) which requires local ablative therapy per Multi-Disciplinary Team (MDT) recommendations) of either:

   (i) Primary NSCLC (Squamous Cell Carcinoma (SCC), Adenocarcinoma, Large Cell) OR (ii) Single pulmonary oligometastatic lesion to be treated for the purpose of the study
6. Patients with central lung tumours/lesions whose radiotherapy plan meets the following criteria:

   (i) OAR eligibility constraints are initially exceeded when full PTV coverage is met; (ii) subsequently meets the CTRIAL-IE 18-33 SOURCE OAR Lung constraints and meets CTRIAL-IE 18-33 SOURCE Lung minimum constraints
7. Inoperable (as per MDT) or patient refuses surgery,
8. Females of childbearing potential must not be pregnant or lactating, must be prepared to take adequate contraception methods during treatment. Males whose female partners are of childbearing potential must be prepared to take adequate contraception methods during treatment. Examples of effective contraception methods are a condom or a diaphragm with spermicidal jelly, or oral, injectable or implanted birth control
9. Absence of psychological, familial, sociological or geographical condition, or psychiatric illness/social situation potentially hampering compliance with the study protocol and follow-up schedule

Exclusion Criteria:

1. Known co-existing or prior malignancy within the last 5 years (except for adequately treated basal cell carcinoma (BCC) or Squamous Cell Carcinoma (SCC) of the skin)) which is likely to interfere with treatment or assessment of outcomes
2. Tumour/oligometastatic lesion that is abutting the oesophagus
3. Evidence of regional (nodal) or distant metastases or metastatic pleural effusion for patients with primary NSCLC
4. Spinal canal involvement
5. Patients with syndromes or conditions associated with increased radiosensitivity
6. Idiopathic pulmonary fibrosis / usual interstitial pneumonia
7. Chemotherapy and/or other targeted therapy administered within 3 months prior to study radiotherapy or planned for <6 weeks following radiotherapy for patients with primary NSCLC, or within 1 week prior to study radiotherapy or planned within 1 week following radiotherapy for patients with an oligometastatic lesion
8. Any previous radiotherapy to the thorax or mediastinum (excluding previous breast or chest wall radiotherapy) which is likely to interfere with treatment or assessment of outcomes
9. Any tumour not clinically definable on the treatment planning CT scan (e.g. surrounding consolidation or atelectasis)
10. Patients unable to undergo 4D-CT scan
11. Uncontrolled intercurrent illness that is likely to interfere with treatment or assessment of outcomes
12. Evidence of any other significant clinical disorder or laboratory finding that makes it undesirable for the patient to participate in the study, or if it is felt by the research / medical team that the patient may not be able to comply with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2020-12-22 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2032-02 (Estimated)

PRIMARY OUTCOMES:
The rate of ≥ Grade 3 treatment-related toxicities occurring between start of treatment and one-year from the end of treatment using NCI CTCAE V5 | From start of treatment to 1 year post treatment
  The rates of ≥ Grade 3 treatment-related adverse events (TxR-AEs) will be calculated as the proportion of evaluable patients (along with the 95% CI) who have any >= Grade 3 treatment-related adverse event occurring between the start of RT and one year post-RT, among the total evaluable patients. These rates will be reported (for applicable patients) by T stage (T1 versus T2 versus T3 versus T4 or combined T stages). The NCI Common Terminology Criteria for Adverse Events (CTCAE Version 5.0) for scoring the treatment-related adverse events will be used.
  The following will be reported at the time of primary endpoint analysis
  * Tabulation of all cases entered, and any patients excluded from the analysis with reasons for exclusion;
  * Distribution of important prognostic baseline and other pre-treatment variables;
  * Frequency and severity of adverse events;
  * Compliance rates of treatment delivery with respect to the protocol prescription

SECONDARY OUTCOMES:
Estimate time to locoregional recurrence/progression, locoregional recurrence-free survival (LRFS), disease-free survival (DFS) and metastasis-free survival rates / further metastasis-free survival rates (for patients with an oligometastatic lesion). | Up to 5 years post treatment
  The Kaplan-Meier method will be used to estimate time to locoregional recurrence; the cumulative proportion surviving without local recurrence at 1- year, 3-years and 5-years; DFS; metastasis-free survival for patients with primary NSCLC; further metastasis-free survival for patients with an oligometastatic lesion. These efficacy endpoints will be expressed as median survival with 95% confidence interval.
Estimates of 1-year, 3-year and 5-year overall survival rates | Up to 5 years post treatment
  The Kaplan-Meier method will be used to estimate time the cumulative proportion surviving (overall survival) at 1-year, 3-years and 5-years.
  Overall survival will be measured from date of registration/ enrolment. Patients alive and free of event at the time of analysis and patients lost to follow-up will be censored at the last available assessment. The event for overall survival is a death due to any cause. The primary time-point of interest is 12 months.

OTHER OUTCOMES:
Post treatment response and outcomes using PET and CT at 3, 6, 9, 12,18, 24, 36, 48 and 60 months post-RT | Up to 60 months (5 years) post treatment
  Only patients who received the prescribed RT dose and who are alive at the specified CT TA timepoints during follow up will be evaluated for tumour response and included in the analysis of tumour response rates. Whole body FDG-PET-CT scan will be done within 18 weeks prior to registration (may be conducted 18-22 weeks prior to registration for some patients, if the patient has had a CT TA within 18 weeks prior to registration), at 6 months and as clinically indicated post-SABR based on review of CT-TA scans.
Acute toxicity profiles on treatment to 3 months post treatment | Up to 3 months post treatment
  Acute toxicity rates will be calculated, summarised and presented in tabular format with proportions plus 95% confidence intervals where appropriate.
Late toxicity profiles to 5 years post treatment | Up to 5 years post treatment
  Late toxicity rates will be calculated, summarised and presented in tabular format with proportions plus 95% confidence intervals where appropriate.
Time to onset of acute and late ≥ Grade 2 and ≥ Grade 3 toxicities | Up to 5 years post treatment
  Time to event will be measured for toxicities (which are related to trial treatment) from treatment start date. Patients alive and free of event at the time of analysis and patients lost to follow-up will be censored at the last available assessment. The primary time-point of interest is 12 months.
Changes in domain-specific Quality of Life (QoL) outcomes at 6 months post treatment compared with outcomes at baseline using the EORTC QLQ C30 (and EORTC QLQ LC13) | From baseline up to 6 months post treatment
  The mean and standard deviation (SD) of the domain-specific EORTC QLQ C30 and EORTC QLQ LC13 scores at baseline and 6 months post treatment will be reported. Scoring will be in line with the published guidelines and will use the QLQ-C30 summary score (excluding financial difficulties and global QOL). The scales are from 1(Not at all) to 4(Very Much) with 1 being the best outcome, and from 1(Very poor) to 7(excellent) with 7 being the best outcome. The proportion of patients who report 'quite a bit' and/or 'very much' for each domain or measure will be reported. Changes in scores over time for each patient will be calculated by subtracting the results at baseline from 6 month results. The mean and SD of the changes will be reported. A Wilcoxon signed rank test will be used to compare differences from baseline. The number of patients who had a clinically meaningful change in QoL as identified by the method recommended by the EORTC QoL Group at the time of analysis will also be reported.
Changes in symptom-specific Quality of Life (QoL) outcomes at 6 months post treatment compared with outcomes at baseline using the EORTC QLQ C30 (and EORTC QLQ LC13) | From baseline up to 6 months post treatment
  The mean and standard deviation (SD) of the symptom-specific EORTC QLQ C30 and EORTC QLQ LC13 scores at baseline and 6 months post treatment will be reported. Scoring will be in line with the published guidelines and will use the QLQ-C30 summary score (excluding financial difficulties and global QOL). The scales are from 1(Not at all) to 4(Very Much) with 1 being the best outcome and from 1(Very poor) to 7(excellent) with 7 being the best outcome. The proportion of patients who report 'quite a bit' and/or 'very much' for each domain or measure will be reported. Changes in scores over time for each patient will be calculated by subtracting the results at baseline from 6 month results. The mean and SD of the changes will be reported. A Wilcoxon signed rank test will be used to compare differences from baseline. The number of patients who had a clinically meaningful change in QoL as identified by the method recommended by the EORTC QoL Group at the time of analysis will also be reported.
Treatment tolerability and feasibility rates based on compliance with prescription and the number of treatment reductions/withdrawals. | Through study treatment, an average of 3 weeks
  Treatment tolerability and feasibility will be measured in terms of the compliance rate for treatment delivery with respect to the protocol prescription and the number of treatment reductions and treatment withdrawals
Pulmonary function changes | Up to 12 months post treatment
  The change in pulmonary function post-treatment will be analysed by calculating the differences in measurements (of PFTs) from baseline to the 12-month follow-up. The descriptive statistics of changes of FEV1 and diffusion capacity before and after treatment will be reported (at least mean, standard deviation, median, and range).
Changes in overall Quality of Life (QoL) outcomes at 6 months post treatment compared with outcomes at baseline using the European Organisation for Research and Treatment of Cancer QoL Questionnaire (EORTC QLQ) C30 and EORTC QLQ Lung Cancer (LC)13 | From baseline up to 6 months post treatment
  The mean and standard deviation (SD) of the overall EORTC QLQ C30 and EORTC QLQ LC13 scores at baseline and 6 months post treatment will be reported. Scoring will be in line with the published guidelines and will use the QLQ-C30 summary score (excluding financial difficulties and global QOL). The scales are from 1 (Not at all) to 4 (Very Much) with 1 being the best outcome, and from 1 (Very poor) to 7 (excellent) with 7 being the best outcome. The proportion of patients who report 'quite a bit' and/or 'very much' for each domain or measure will be reported. Changes in scores over time for each patient will be calculated by subtracting the results at baseline from 6month results. The mean and SD of the changes will be reported. A Wilcoxon signed rank test will be used to compare differences from baseline. The number of patients who had a clinically meaningful change in QoL as identified by the method recommended by the EORTC QoL Group at the time of analysis will also be reported.
Develop a platform for prediction and monitoring of treatment response/toxicities using Raman spectra of the cellular and plasma fraction of the patient blood. (Sub-Study 1) | 9 months follow-up
  Raman spectra will be recorded from both lymphocytes and plasma to produce a library of spectral measurements in patients pre- and post-treatment. Advanced multivariate and machine learning methodologies will be used to develop a platform for prediction and monitoring of treatment response/toxicities using Raman spectra of the cellular and plasma fraction of the patient blood.
Identify blood biomarkers as indicators for toxicity/relapse and the development of a panel of predictive/prognostic biomarkers. (Sub-Study 2) | 9 months follow up
  To detect changes in protein expression profiles that may predict outcome and identify prognostic biochemical markers of early toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Prof. John Armstrong, MD FRCPI DABR FFRRCSI, Principal Investigator — Cancer Trials Ireland/ St Luke's Radiation Oncology Network
Locations (2):
- Ireland (2):
  - Beacon Hospital, Dublin
  - St Luke's Radiation Oncology Network (SLRON) at St Luke's Hospital and St James's Hospital, Dublin

IPD SHARING:
Plan to Share IPD: Undecided